CLINICAL TRIAL: NCT05265429
Title: Biology of Young Lung Cancer Study: The YOUNG LUNG Study
Status: Recruiting | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Pasi Janne, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 21-442
Record Dates: First submitted 2022-02-16; First posted 2022-03-03 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Non Small Cell Lung Cancer; Small Cell Lung Carcinoma; NUT Carcinoma
Keywords: Non Small Cell Lung Cancer; Small Cell Lung Carcinoma; Genetics; Genomics; Young lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — whole blood, serum, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Data/Biospecimen Collection: Tumor and saliva specimens from participants with non-small cell lung cancer (NSCLC) or small cell lung cancer (SCLC) diagnosed at age 45 or younger
  Interventions: Genetic: Data and Specimen Collection

INTERVENTIONS:
Genetic: Data and Specimen Collection — * Provide research team access to relevant medical records
  * Answer two (2) short questionnaires at time of consent
  * Provide up to 5 tubes (37 ml) of blood at or near the time of consent, and/or saliva sample
  * Consider consenting to other optional parts of the research such as:
    * Providing additional blood or tissue samples in the future (optional)
    * Providing permission for obtainment of stored tissue specimens from lung cancer surgeries or biopsies from the pathology departments where they have been stored (optional)

SUMMARY:
The purpose of this research study is to learn more about lung cancer (NSCLC or SCLC) diagnosed in adults at ages 45 or younger.

DETAILED DESCRIPTION:
This research study looks to enroll as many people diagnosed with lung cancer at 45 years old or younger in order to:

* Better understand causes of lung cancer in individuals 45 years old and younger, which is a rare disease
* Better estimate lung cancer risks and potential risk factors for lung cancer in individuals 45 years old and younger
* Examine tumor (somatic) or normal (germline) genetic changes that may be shared among young lung cancer patients
* Improve opportunities for screening and treatment of lung cancer in individuals 45 years old and younger

Study procedures will include:

* Collecting information from participants' medical record and two (2) short questionnaires
* Collecting blood and/or saliva samples
* Collecting tumor tissue samples (optional)

It is expected that about 500 people will take part in this research study. Participants will be in this study until it closes or the participant withdraws consent.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 and under at lung cancer diagnosis
* Pathologically confirmed bronchogenic lung carcinoma (NSCLC or SCLC of any stage) at any treatment time point
* Provision of written informed consent
* Willingness to undergo no more than two (2) peripheral blood draws in a four (4) week period, with no more than 50 ml peripheral blood collected over eight (8) weeks
* Individuals under age 18 are eligible for study if they meet defined criteria; in addition, consent for participation must be given by a legal guardian or parent

Exclusion Criteria:

* Individuals who decline to sign consent
* Individuals who are unable to give consent or assent and are without a designated healthcare proxy
* Compromise of patient diagnosis or staging if tissue is used for research

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults age 45 or under at time of non-small lung cancer (NSCLC) or small cell lung cancer (SCLC) diagnosis
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Repository of specimens and data | 5 years or study closure
  Prospective registry of young lung cancer specimens for exploratory tumor and germline genomics, transcriptomics/proteomics, and future biomarker study.

SECONDARY OUTCOMES:
Number of patients with targetable somatic alterations in known oncogenic driver genes | 5 years or study closure
  Targetable alterations are defined as any somatic alteration in a driver oncogene for which a Food and Drug Administration-approved therapy exists, for which an off-label therapy exists, or for which a clinical trial exists (including but not limited to EGFR, KRAS, ALK, ROS1, RET, MET, BRAF, and TRK). Results will be summarized using descriptive statistics.
Number of patients with predicted oncogenic alterations in unknown driver genes | 5 years or study closure
  Unknown driver genes include genes not currently known to be driver oncogenes in lung cancer, and for which no directed treatment exists. Results will be summarized using descriptive statistics.
Number of patients with pathogenic or likely pathogenic germline alterations in known cancer predisposition genes | 5 years or study closure
  Pathogenic or likely pathogenic variants based on classification by the American College of Medical Genetics and Genomics (ACMG). Results will be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Pasi A Janne, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu